CLINICAL TRIAL: NCT06195618
Title: ESTUDIO CLÍNICO FASE I DE INMUNOTERAPIA CON VACUNAS SINTÉTICAS PERSONALIZADAS EN PACIENTES CON CÁNCER DE MAMA TRIPLE NEGATIVO
Brief Title: Personalized Vaccine for TNBC Immunotherapy
Acronym: TEBICA003 TNBC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Fundación Salud de los Andes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEBICA003
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Female
Keywords: Triple negative breast cancer; Neo-adjuvant chemotherapy; Dendritic cells; Peptide; Immunotherapy; Immune-monitoring; Personalized vaccines
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccine (Experimental): Triple-negative breast cancer patients with specific tumor mutation, with six doses of peptide-pulsed autologous dendritic cells after surgery
  Interventions: Biological: Peptide (neoantigen) pulsed autologous Dendritic cell

INTERVENTIONS:
Biological: Peptide (neoantigen) pulsed autologous Dendritic cell — Intradermal vaccination with peptide-pulsed autologous dendritic cells in 200 µL of patient's serum in six doses, one weekly after surgery.

SUMMARY:
Due to their genetic instability, breast tumors that do not express receptors for Estrogens, Progestagens or amplify the Her2 / neu oncogene [called triple-negative breast cancer (TNBC)] and other tumors such as melanoma, non-small cell lung cancer, accumulate numerous mutations that make them highly resistant to different regimens of chemo- or radiotherapy, thereby generating high morbidity and mortality. However, immunology can turn the genetic instability of tumors into the Achilles' tendon. Evidence of this has been revealed in Phase I clinical studies in patients with melanoma and lung cancer in an advanced stage of metastasis treated with Ipilimumab (anti-CTLA4) to decrease immunosuppression, in whom peptides containing mutations presented in Major Complex molecules Histocompatibility of Class I (MHC I) of the tumor itself results in their recognition as "foreign" neo-antigens leading to the efficient destruction of the tumor by anti-tumor CD8 + T lymphocytes that are amplified when they are vaccinated with these peptides.

For this reason, the identification of non-synonymous mutations of single amino acid and vaccination with 25 amino acid peptides that incorporate these mutations (synthetic vaccines) is emerging today as an alternative for immunotherapy of cancers responsible for high mortality in humans. In an approach that takes 16 weeks, today, it is possible to go from the analysis of the tumor's transcriptome (which allows identifying the universe of tumor mutations) to the patient's vaccination with a personalized vaccine that contains neo-antigens of his tumor.

TNBC is the most aggressive breast tumor, representing around 15% of breast cancers in our environment. While generally, at least 30% of women with other types of metastatic breast cancer survive 5 years after diagnosis, most patients diagnosed with metastatic TNBC die within this time. The lack of selective therapies and the poor prognosis of patients with TNBC make their therapeutic management difficult, so the implementation of new therapies for this type of tumor is the main focus of researchers who seek more effective and selective treatments to improve the life expectancy of patients without compromising their quality of life. The genetic instability and high rate of mutations of the TNBC most likely favor the generation of neo-epitopes. Still, due to the immunosuppressive environment of the tumor, it escapes the immunosurveillance of the immune system. Despite the high mortality induced by this tumor, a percentage of patients treated with neoadjuvant chemotherapy with agents such as Doxorubicin and Cyclophosphamide (AC) + Taxanes respond to this chemotherapy regimen. In particular, the anti-tumor effect of AC is attributed to two things: (i) the direct cytotoxic effect on the tumor cell, (ii) the immunostimulation of T lymphocytes promoted by Immunogenic Cell Death (ICD) selectively induced by these drugs. Therefore, in this project, we propose to carry out the first clinical study in Colombia of vaccination of patients with TNBC with synthetic peptides that contain mutations of their own tumor to evaluate the immunogenicity and safety of this type of personalized vaccine as a therapeutic alternative for this tumor. Achieving the specific objectives set out in this project would mean that we have been validated in Colombia the experimental design necessary to identify unique epitopes in tumors and demonstrate the safety and immunogenicity of these vaccines. We consider that having achieved the above; we will have taken an important step towards the implementation in our country of the use of this type of vaccine for immunotherapy not only of TNBC but of other tumors such as glioblastoma, gastric, esophagus, and pancreas, highly fatal due to its high mutation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 75 years of age.
2. Histologically confirmed diagnosis of primary triple negative breast carcinoma (TNBC).
3. Patients who have already been treated, either with chemo/radiotherapy and/or surgery regimens, and in whom, according to previous preclinical studies, it was possible to clearly identify tumor NEOANTIGENS expressed by their tumor.
4. Have frank venous access.
5. Have a functional status (Karnofsky Scale) greater than 70%.
6. Weight equal to or greater than 50 kilograms.
7. The chemical synthesis of at least one tumor NEOANTIGEN expressed exclusively by your tumor was successful.
8. The apheresis procedure successfully allowed the obtaining of sufficient white blood cells to obtain leukocytes necessary for functional tests and for the derivation of dendritic cells.

Exclusion Criteria:

1. Active and/or uncontrolled cardiovascular disease.
2. You are pregnant or breastfeeding.
3. Has associated medical comorbidities such as diabetes or kidney failure, or coagulation disorders.
4. You have been hospitalized in the last month.
5. Has another active primary tumor except for skin tumors.
6. Patients who are linked to another clinical study.
7. Patients with a history of infectious diseases such as HIV, Hepatitis, tuberculosis.
8. Consumption of immunosuppressive medications such as corticosteroids (except topical).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse effects | From day 0 (vaccination 1) until 3 month after last vaccination
  Evaluation of number and severity of the adverse effects in the vaccinated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina - Universidad Nacional de Colombia, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernal-Estevez DA, Ortiz Barbosa MA, Ortiz-Montero P, Cifuentes C, Sanchez R, Parra-Lopez CA. Autologous Dendritic Cells in Combination With Chemotherapy Restore Responsiveness of T Cells in Breast Cancer Patients: A Single-Arm Phase I/II Trial. Front Immunol. 2021 Aug 20;12:669965. doi: 10.3389/fimmu.2021.669965. eCollection 2021. PMID 34489928